CLINICAL TRIAL: NCT04385459
Title: Long Term Follow-up (=> 5 Years) for Transcatheter Aortic Valve Implantation in Patients With Severe Aortic Valve Stenosis and Concomitant Coronary Artery Disease
Brief Title: Severe Aortic Valve Stenosis and Concomitant Coronary Artery Disease in Patients Undergoing TAVI
Status: Completed | Type: Observational
Sponsor: Örebro County Council (Other Government)
Responsible Party: Principal Investigator, Ninos Samano M.D., MD, PhD, Örebro County Council
Other Study IDs: 273468
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2021-09-09 (Actual); Status verified 2021-09

CONDITIONS: Aortic Valve Stenosis; Coronary Artery Disease
Keywords: Aortic valve stenosis; Coronary artery disease; Transcatheter aortic valve implantation; Mortality
MeSH Terms: conditions — Aortic Valve Stenosis; Coronary Artery Disease | interventions — JCAD protein, mouse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients without coronary artery disease: No prior coronary intervention and no significant stenosis noted during coronary angiography.
- Patients with coronary artery disease: Our definition of coronary artery disease is:
  * Prior coronary artery bypass grafting or percutaneous coronary intervention
  * Significant stenosis or occlusion noted during coronary angiography
  Interventions: Other: Coronary artery disease

INTERVENTIONS:
Other: Coronary artery disease — Exposure
  Groups: Patients with coronary artery disease

SUMMARY:
Patients undergoing surgical aortic valve replacement (sAVR) with concomitant coronary artery disease (CAD) are known to have higher mortality rates compared to patients without CAD. This same phenomenom has not been clearly mapped in patients with CAD that goes through a transcatheter aortic valve implantation procedure.

DETAILED DESCRIPTION:
A narrowing of the aortic valve, aortic stenosis, is a relatively common condition among the elderly. When the narrowing gets too severe, symptoms such as loss of breath, angina and fainting can occur, so called symptomatic aortic stenosis. Since the 60's, surgical aortic valve replacement (sAVR) has been the treatment of choice for severe aortic stenosis. A large setback of this method is that a third of these patients could not undergo the treatment due to too high surgical risk.

Transcatheter aortic valve implantation (TAVI) have steadily gained ground in the treatment of severe aortic valve stenosis during the last decade. The procedure, which is a minimal invasive type of surgery, introduces a new aortic valve through a catheter, usually transfemorally. Patients with an underlying coronary artery disease (CAD) undergoing sAVR is known to have higher mortality rates postoperatively. However, it is not clearly known how an underlying CAD affects the long term results after a TAVI-surgery. It is therefore our goal to contribute with the mapping of how a CAD affects the long term results for patients with a severe aortic valve stenosis that undergoes TAVI.

ELIGIBILITY:
Inclusion Criteria:

* All patients that underwent a TAVI procedure at Örebro University Hospital between 2009 till 1st december 2019.

Exclusion Criteria:

* Patients with procedural-related coronary artery injury and patients with solitary stenosis in a diagonal branch were excluded from the study.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients that underwent a TAVI procedure at Örebro University Hospital between the time period 2009 till 1st december 2019 were included.
Sampling Method: Probability Sample
Enrollment: 346 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-12-24 (Actual); Study Completion 2020-12-24 (Actual)

PRIMARY OUTCOMES:
Mortality | Five years.
  Death after the procedure

SECONDARY OUTCOMES:
Factors associated with less favorable early and late mortality | Five years
  Factors such as renal function or comorbidities associated with higher mortality.

CONTACTS AND LOCATIONS:
Overall Officials: Ninos Samano, MD,PhD, Principal Investigator — Department of Cardiothoracic and Vascular Surgery, Örebro University
Locations (1):
- Department for Cardiothoracic and Vascular Surgery, Örebro University Hospital, Örebro, Sweden